CLINICAL TRIAL: NCT07308743
Title: Impact of Computer-aided Detection System on the Proximal Adenoma Miss Rate: a Multicenter Tandem Rondomized Controlled Trial
Brief Title: Impact of Computer-aided Detection System on the Proximal Adenoma Miss Rate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: The Fifth Affiliated Hospital of Zunyi Medical College (Other); Longgang District People's Hospital of Shenzhen (Other); Yangjiang People's Hospital (Other); Jiangmen Central Hospital (Other); Dongguan Shuixiang Central Hospital (Unknown); Pingshan District People's Hospital of shenzhen (Unknown); Huizhou Third People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NFEC-2025-679
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Colon Adenomas; Colon Polyps; Sessile Serrated Lesion
Keywords: computer-aided detection; proximal adenoma miss rate; Randomized Tandem Colonoscopy Study
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Prospective randomized design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-aided detection-assisted colonoscopy (Experimental): Tandem colonoscopy of proximal colon assisted with computer-aided detection system followed by conventional white-light colonoscopy
  Interventions: Device: Computer-aided detection-assisted colonoscopy
- Conventional white-light colonoscopy (Active Comparator): Tandem conventional white-light colonoscopy of proximal colon followed by usual computer-aided detection-assisted colonoscopy
  Interventions: Procedure: Conventional white-light colonoscopy

INTERVENTIONS:
Device: Computer-aided detection-assisted colonoscopy — Computer-aided detection-assisted colonoscopy for detection of colonic polyp
  Arms: Computer-aided detection-assisted colonoscopy
Procedure: Conventional white-light colonoscopy — Conventional white-light colonoscopy
  Arms: Conventional white-light colonoscopy

SUMMARY:
This is a prospective, multicenter randomized controlled trial designed to determine whether the use of computer-aided detection system could reduce the miss rates of adenomas, SSLs, and polyps in the proximal colon during tandem colonoscopy.

DETAILED DESCRIPTION:
1. Study Centers 1) Nanfang Hospital, Southern Medical Univerisity, Guangzhou, China 2) The Fifth Affiliated Hospital of Zunyi Medical University, Zhuhai, China 3) Longgang District People's Hospital of Shenzhen, Shenzhen, China 4) Yangjiang People's Hospital, Yangjiang, China 5) Jiangmen Central Hospital, Jiangmen, China 6) Huizhou Third People's Hospital, Huizhou, China 7) Dongguan Shuixiang Central Hospital, Dongguang, China 8) Pingshan District People's Hospital of Shenzhen, Shenzhen, China
2. Study population 1) Inclusion criteria:

   1. Patients age 40-75 years old, regardless of gender
   2. Patients presenting for physical examination, colorectal cancer screening or diagnosis
   3. Patients voluntarily signs an informed consent form 2) Exclusion criteria:

   <!-- -->

   1. Unable to cooperate ot tolerate colonoscopy
   2. History of inflammatory bowel disease
   3. History of colorectal cancer
   4. Previous colorectal surgery
   5. History of recurrent constipation
   6. Taking anticoagulant and antiplatelet drugs berfore procedure
   7. High risk conditions such as severe cardiovascular and cerebrovascular diseases, severe anemia, or uncorrected infections
   8. Pregnant or lactating women Researchers concluded that patient was not suitable to participate in this trial.

      3) Post-randomization exclusion criteria:

   <!-- -->

   1. Cecum could not be intubated for various reasons
   2. Boston Bowel Preparation Scale (BBPS) score of the proximal colon is <2
3. Study design This is a prospective , multicenter randomized controlled trial comparing the miss rates of proximal colonic lesions (including adenomas, SSLs, and polyps) by computer-aided detection-assisted colonoscopy or conventional colonoscopy. The study will be conducted in the Endoscopy Centre of the participating hospitals.
4. Randomization 1) Eligible patients at each center will be randomized (1:1) to computer-aided detection-assisted colonoscopy first or conventional white light colonoscopy first, followed immediately by the other procedure in tandem fashion by the same endoscopist. The proximal colon is defined as the colonic segment proximal to the hepatic flexure.

2) Randomization will be performed using computer-generated random sequences in blocks of 6, with stratification by academic level of participation center, experience of endoscopists, and indications of colonoscopy. Patients will be blinded to their group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 40-75 years old, regardless of gender
2. Patients presenting for physical examination, colorectal cancer screening or diagnosis
3. Patients voluntarily signs an informed consent form

Exclusion Criteria:

1. Unable to cooperate ot tolerate colonoscopy
2. History of inflammatory bowel disease
3. History of colorectal cancer
4. Previous colorectal surgery
5. History of recurrent constipation
6. Taking anticoagulant and antiplatelet drugs berfore procedure
7. High risk conditions such as severe cardiovascular and cerebrovascular diseases, severe anemia, or uncorrected infections
8. Pregnant or lactating women Researchers concluded that patient was not suitable to participate in this trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proximal adenoma missed rate | One day
  The number of adenomas identified during the second right colon inspection divided by the overall number of adenomas identified during the first and second right colon inspection.

SECONDARY OUTCOMES:
Proximal polyp missed rate | One day
  The number of polyps identified during the second right colon inspection divided by the overall number of polyps identified during the first and second right colon inspection.
Proximal SSLs missed rate | One days
  The number of SSLs identified during the second right colon inspection divided by the overall number of SSLs identified during the first and second right colon inspection.
Proximal advanced adenoma missed rate | One day
  The number of advanced adenomas identified during the second right colon inspection divided by the overall number of advanced adenomas identified during the first and second right colon inspection.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided